CLINICAL TRIAL: NCT01629368
Title: A Single-Center, Open-Label, One-Sequence, Crossover Study to Investigate the Effects of Multiple Doses of Carbamazepine on the Pharmacokinetics of a Single Dose RO4917523 in Healthy Subjects
Brief Title: A Study of the Effect of Carbamazepine on the Pharmacokinetics of RO4917523 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: BP28256; 2012-000771-16 (EudraCT Number)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Carbamazepine; 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

ARMS (2):
- Dosing Period 1 (Experimental)
  Interventions: Drug: RO4917523
- Dosing Period 2 (Experimental)
  Interventions: Drug: Carbamazepine; Drug: RO4917523

INTERVENTIONS:
Drug: Carbamazepine — Multiple doses of carbamazepine
  Arms: Dosing Period 2
Drug: RO4917523 — Single dose of RO4917523

SUMMARY:
This single-center, open-label, cross-over study will evaluate the effect of carbamazepine on the pharmacokinetics of RO4917523 in healthy volunteers. Healthy volunteers will receive a single dose of RO4917523 alone and in combination with multiple doses of carbamazepine in a cross-over design. The anticipated time on study treatment is 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18-65 years of age inclusive
* Non-smokers
* Body mass index (BMI) between 18 and 30 mg/m2 inclusive
* Women who are not menopausal or surgically sterile agree to use two adequate methods of contraception

Exclusion Criteria:

* Evidence of any active or chronic disease
* History of any significant disease (e.g., cardiovascular, hepatic, renal) or cancer
* History or presence of clinically significant psychiatric condition
* Any condition or disease that would render the volunteer unsuitable for the study, place the volunteer at undue risk or interfere with the ability of the volunteer to complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration time curve | Period 1: Pre-dose and up to Day 14, Period 2: Pre-dose and up to Day 29

SECONDARY OUTCOMES:
Safety: incidence of adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France